CLINICAL TRIAL: NCT01664520
Title: The Effects of Dexmedetomidine on Cerebral Autoregulation and Cerebral Oxygenation in Subarachnoid Haemorrhage Patients
Brief Title: Dexmedetomidine and Subarachnoid Haemorrhage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Riikka Takala, MD, PhD Senior Staff Anaesthesiologist, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Turku University Hospital; 2012-000068-11 (EudraCT Number); KLNRO 45/2012 (Other: Finnish Medicines Agency)
Record Dates: First submitted 2012-08-04; First posted 2012-08-14 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Subarachnoid Hemorrhage; Aneurysm
Keywords: Subarachnoid hemorrhage; Dexmedetomidine; Autoregulation; Intracranial pressure; Cerebral oxygenation
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomine infusion (Experimental)
  Interventions: Drug: Dexmedetomidine infusion

INTERVENTIONS:
Drug: Dexmedetomidine infusion — Both static and dynamic autoregulation are assessed first during propofol infusion, before commencement of dexmedetomidine infusion. Dexmedetomidine infusion is commenced with a dose of 0.7 μg/kg/h and propofol infusion is stopped concomitantly. After 2 hours dexmedetomidine infusion, the static and dynamic autoregulation are assessed. If there are no signs of worsening of autoregulation, then the dexmedetomidine infusion is increased to 1 μg/kg/h and after 2 hours the static and dynamic autoregulation are assessed again. However, if autoregulation worsens during dexmedetomidine infusion, it will be stopped and further testing with dexmedetomidine will not be carried out. If autoregulation does not worsen with the 1 μg/kg/h dose then the dose will be increased to 1.4 μg/kg/h. After 2 hours infusion the dynamic and static autoregulation are assessed again.
  Blood samples for determining dexmedetomidine plasma concentration are collected alongside with the autoregulation assessments

SUMMARY:
The purpose of this study is to investigate how dexmedetomidine affects static and dynamic autoregulation, intracranial pressure (ICP) and cerebral oxygenation in aneurysmal subarachnoid haemorrhage (SAH) patients.

DETAILED DESCRIPTION:
Dexmedetomidine is a selective α2-agonist which induces sedation, anxiolysis and analgesia without respiratory depression. These effects, as well as neuroprotective properties in experimental studies would be ideal in neuroanaesthesia and in neurocritical care. Poor grade SAH patients are treated in intensive care units (ICU). These patients are sedated often with propofol. However, to assess the patient's neurology, the propofol sedation must be stopped and the wakening of the patient may take time. Dexmedetomidine would be more advantageous, allowing wakening during the infusion. However, the effects of dexmedetomidine on cerebral autoregulation are unknown in SAH patients.

15 SAH patients requiring sedation, mechanical ventilation and ICP monitoring will be rolled in to the study.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal SAH
* Aneurysm treated with coil(s) or clip(s)
* Age 18-80 years
* Written informed consent from the next of kin

Exclusion Criteria:

* Pregnancy
* Nursing woman
* Sick sinus syndrome
* Carotid stenosis
* Heart rate less than 50 beats / minute
* Mean arterial pressure less than 50 mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Change in autoregulation, ICP and cerebral oxygenation | 2, 4 and 6 hours
  Autoregulation is assessed using transcranial doppler (TCD) and ICP amplitude analysis. ICP and cerebral oxygenation are part of standard multimodal monitoring and these are continuously monitored and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Riikka SK Takala, MD PhD, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland